CLINICAL TRIAL: NCT04981587
Title: Effects of Strength Exercise on Fall Risk in Elderly With Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIH/FEB.21/8.TES
Record Dates: First submitted 2021-07-19; First posted 2021-07-29 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Disease; Dementia; Alzheimer's Type (Etiology); Fall Risk; Elderly; Resistance Training
Keywords: alzheimer disease; elderly; exercise; fall risk
MeSH Terms: conditions — Alzheimer Disease; Dementia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This is the group that receives strength exercise in addition to usual treatment
  Interventions: Procedure: Strength exercise; Other: Usual treatment
- Control group (Other): This is the group that only receives usual treatment
  Interventions: Other: Usual treatment

INTERVENTIONS:
Procedure: Strength exercise — Strength exercise protocol for upper and lower limbs, using weights and elastic bands
  Arms: Intervention group
Other: Usual treatment — The usual treatment is based on activities to enhance brain functions: attention, memory, executive functions, language and orientation.

SUMMARY:
Interventional study to show the effects of strength exercise on fall risk in elderly with Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

* accept to participate in the study, through informed consent
* subjects aged 60 or over with medical diagnosis of Azlheimer´s disease
* minimal physical and mental state to perform the cognitive tests and strength exercise routine

Exclusion Criteria:

* Neurodegenerative disease other than Alzheimer's disease
* Suffering from serious somatic or psychiatric illnesses
* Patients who have practiced strength exercise regularly

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline Short physical performance battery (SPPB) at 3 and 6 months | Baseline, 3 and 6 months (3 months after intervention)
  Informs about fall risk and mobility Score: 0-12 High score means better result

SECONDARY OUTCOMES:
Change from baseline Activities specific balance confidence scale (ABC scale) at 3 and 6 months | Baseline, 3 and 6 months (3 months after intervention)
  This questionnaire allows to measure the balance of a person Score: 0-100% High percentage means better result
Change from baseline Lawton Instrumental Activities of Daily Living Scale (IADL) at 3 and 6 months | Baseline, 3 and 6 months (3 months after intervention)
  This tool gives us information about performance in activities of daily living Score: 0-8 High score means better result
Change from baseline Quality of life Alzheimer Disease (QoL-AD) at 3 and 6 months | Baseline, 3 and 6 months (3 months after intervention)
  Through this test we can know the level of quality of life of users who suffer from this disease Score: 0-52 High score means better result
Change from baseline FRAIL test at 3 and 6 months | Baseline, 3 and 6 months (3 months after intervention)
  This rapid test allows to determine the state of frailty of older people Score: 0-5 High score means worst result
Change from baseline Mini Mental State Examination (MMSE) at 3 and 6 months | Baseline, 3 and 6 months (3 months after intervention)
  This test gives us information about the cognitive performance of the participants Score: 0-30 High score means better result
Change from baseline Neuropsychiatric Inventory (NPI-Q) at 3 and 6 months | Baseline, 3 and 6 months (3 months after intervention)
  This tool allows to specify the neuropsychiatric symptoms patients present Score: 0-36 High score means worst result
Change from baseline Manual dynamometry at 1,2,3 and 6 months | Baseline, 1, 2, 3 and 6 months (3 months after intervention)
  This test allows to quantify force an individual presents in a simple way Score: 0-∞ High score means better result
Modified Borg scale | 3 times/week during strength exercises sessions
  In this way we can measure the level of perceived exertion during the intervention with strength exercise Score: 0-10 High score means more fatigue
Change from baseline One Maximum repetition strength test (1 MR) at 1,2,3 and 6 months | Baseline, 1 , 2 , 3 and 6 months (3 months after intervention)
  Allows you easily to assess maximum strength Score: 0-∞ High score means more strength level

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Achalandabaso, Phd, Study Director — University of Jaen
Locations (2):
- Spain (2):
  - A.F.A La Estrella, Jaén, Andalusia
  - Alexander achalandabaso, Alcalá de Henares, Madrid